CLINICAL TRIAL: NCT06358482
Title: Electric Toothbrush Efficacy in Preventing Dental Plaque Development: A RCT Using QLF Technology
Brief Title: Electric Toothbrush Efficacy in Preventing Dental Plaque Development
Acronym: E-TOOTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riccardo Polosa (Other)
Responsible Party: Sponsor-Investigator, Riccardo Polosa, Full Professor, Universita degli Studi di Catania
Organization: Universita degli Studi di Catania (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORAL1
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Dental Plaque; Calculus, Dental
MeSH Terms: conditions — Dental Plaque; Dental Calculus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A Digital (Experimental): oscillating-rotating electric toothbrush group
  Interventions: Behavioral: oscillating toothbrush
- B Manual (Active Comparator): manual toothbrush group
  Interventions: Behavioral: standard manual toothbrush

INTERVENTIONS:
Behavioral: oscillating toothbrush — oscillating toothbrush
  Arms: A Digital
Behavioral: standard manual toothbrush — standard manual toothbrush
  Arms: B Manual

SUMMARY:
The present study will be the first to compared dental plaque quantitation between an oscillating-rotating electric toothbrush and a manual toothbrush with a new QLF technology.

DETAILED DESCRIPTION:
This is a randomized controlled trial of 12-weeks duration designed to assess whether a new commercially available oscillating-rotating electric toothbrush can objectively improve dental plaque parameters obtained via light induced fluorescence (QLF) technology. The study will be conducted in a dental clinic in Italy

ELIGIBILITY:
Inclusion Criteria:

* healthy adult (aged 18-50 years)
* non-smokers
* without clinical signs of periodontitis with at least 10 natural anterior teeth in total (cuspid to cuspid and lower and upper jaw).

Exclusion Criteria:

* significant oral soft tissue pathology or any type of gingival overgrowth other than plaque-induced gingivitis,
* with fixed and removable orthodontic appliances or removable dentures,
* with any other medical condition that, in the opinion of the principal investigator, would jeopardize the participant's safety or diminish the validity of study results

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
fluorescence intensity of at least 30% (ΔR30) | 120 DAYS
  1) the percentage of the total tooth surface showing an increase in the fluorescence intensity of at least 30% (ΔR30) - this indicates the total area of mature dental plaque detected,
the fluorescence intensity of at least 120% (ΔR120) | 120 DAYS
  2) the percentage of the total tooth surface showing an increase in the fluorescence intensity of at least 120% (ΔR120) - this reveals just areas of greater level of plaque thickness/maturation (i.e. calculus/tartar) within the total area of mature dental plaque detected.

SECONDARY OUTCOMES:
oral hygiene (SOH) scoring, The score can be from 0, 1, .. to 5. A SOH value of 0 indicates no plaque, and 5 is the maximum and stands for maximum plaque teeth coverage an is the worst state. | 120 DAYS
  3) the simple oral hygiene (SOH) scoring - this score is calculated by the proprietary software and provides an estimate of the degree of gingival inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- ADDENDO, Catania, Italy

IPD SHARING:
Plan to Share IPD: No